CLINICAL TRIAL: NCT04080128
Title: Examination of Myopia Progression and Consequences and Mechanisms of Soft Bifocal Contact Lens Myopia Control
Brief Title: Examination of Myopia Progression and Soft Bifocal Contact Lens Myopia Control
Acronym: BLINK2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Houston (Other)
Responsible Party: Principal Investigator, Jeffrey J. Walline, OD PhD, Principal Investigator, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UG1EY023206 (NIH)
Record Dates: First submitted 2019-08-27; First posted 2019-09-06 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Contact lens (Other): Depending upon the study lens proven to be the most effective in the BLINK Study, this contact lens will be used for the first two years of the study. The last year of the study, all subjects will be wearing single vision contact lenses.
  Interventions: Device: Contact lenses

INTERVENTIONS:
Device: Contact lenses — Depending on the results of the BLINK Study either a single vision spherical contact lens or a multifocal contact lens.

SUMMARY:
This project intends to provide important, previously unmet answers regarding biological associations with myopia (nearsightedness) progression in order to improve the ability to predict patients who are most likely to benefit from myopia control, as well as questions frequently posed by patients and practitioners about the side effects, mechanism, and discontinuation of soft bifocal contact lens myopia control. The first three aims examine the association between biological variables that can be measured non-invasively and myopia progression, and they will be conducted regardless of the outcome of the currently in progress BLINK Study. The last three specific aims will be conducted if soft bifocal contact lenses slowed myopia progression by 30% or more in the BLINK Study, and they can be investigated with very few additional measurements.

DETAILED DESCRIPTION:
The primary goal of the BLINK2 Study is to determine correlates of myopia progression using non-invasive measurement of biomarkers, such as choroidal thickness and intrinsically photosensitive retinal ganglion cell-mediated pupil function, and outdoor light exposure in children. If multifocal contact lenses slow the progression of myopia by 30 percent or more compared to single vision contact lenses during the BLINK Study, the investigators will also answer important questions about the consequences and mechanism of the treatment effect, such as whether multifocal contact lens wear alters accommodative function and whether or not the treatment benefit is transient. Specifically, the investigators will investigate whether myopia progression is slowed or simply delayed by multifocal contact lens wear and whether there is a rebound in myopia progression, an increase in progression rate, after discontinuation of multifocal contact lenses. The investigators will identify myopic children who will most benefit from myopia control by determining those who are most likely to progress, thereby maximizing the potential for benefit and minimizing risk. The investigators will accomplish this goal by investigating the effect on progression of the most important ocular and environmental risk factors recently hypothesized to control eye growth. The project will collect the most extensive longitudinal dataset ever on choroidal thickness in childhood myopia. The investigators will test the important question of whether time outdoors and light exposure influence myopia progression after onset in addition to whether these affects are mediated by intrinsically photosensitive retinal ganglion cells. If soft multifocal contact lenses show a clinically meaningful slowing of myopia progression, we will also answer important questions asked routinely by our clinical colleagues. The investigators will know the accommodative effect of multiple years of multifocal contact lens wear in children, the investigators will know if multifocal contact lenses slow or simply delay myopia progression, and the investigators will know whether myopia progression increases following discontinuation of soft multifocal contact lens wear. Answers to questions addressed by this proposal could improve care for 60 million myopic children in the United States. While the consequences of ordinary myopia are rarely sight-threatening, the quality of life for myopic patients is negatively affected and the health care costs to treat myopia are approximately 4.6 billion dollars in 1990 US dollars. The National Eye Institute recognizes the need to evaluate the efficacy of potential treatments for delaying the onset or for slowing the progression of myopia, such as lenses that alter peripheral defocus. The BLINK2 Study seeks to maximize benefit while lowering the risk of multifocal contact lens wear for myopia control while answering important scientific and clinical questions about the consequences and mechanism of myopia progression, a problem that affects many people in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the BLINK Study

Exclusion Criteria:

-

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 248 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
The statistical correlation between choroidal thickness and axial length | Three years
  test the hypothesis that thinner subfoveal choroidal thickness (a layer of blood vessels) is associated with greater axial elongation (eye growth)
The statistical correlation between iPRGC activity and axial length | Three years
  test the hypothesis that less ipRGC activity (cells in the back of the eye as measured by blue light-driven inputs to the pupil response) is associated with greater axial elongation (eye growth)
The statistical correlation between Light levels and axial length | Three years
  test the hypothesis that exposure to lower light levels is associated with greater axial elongation (eye growth)

SECONDARY OUTCOMES:
Accommodative amplitude | Two years
  In the event of an effect of multifocal contact lens on myopia progression, the investigators will test the hypothesis that long-term soft bifocal contact lens wear does not alter accommodative amplitude. This hypothesis predicts that at the baseline BLINK2 Study visit, the accommodative amplitude will be similar across the three treatment groups that were randomly assigned at the beginning of the BLINK Study; if they are not similar, they will become similar over the next two years.
Lag of accommodation | Two years
  In the event of an effect of multifocal contact lens on myopia progression, the investigators will test the hypothesis that long-term soft bifocal contact lens wear does not alter accommodative lag. This hypothesis predicts that at the baseline BLINK2 Study visit, accommodative lag will be similar across the three treatment groups that were randomly assigned at the beginning of the BLINK Study; if they are not similar, they will become similar over the next two years.
Accommodative facility | Two years
  In the event of an effect of multifocal contact lens on myopia progression, the investigators will test the hypothesis that long-term soft bifocal contact lens wear does not alter accommodative facility. This hypothesis predicts that at the baseline BLINK2 Study visit, the accommodative facility will be similar across the three treatment groups that were randomly assigned at the beginning of the BLINK Study; if they are not similar, they will become similar over the next two years.
Slowing of myopia progression | Two years
  In the event of an effect of multifocal contact lens on myopia progression, the investigators will test the hypothesis that soft bifocal contact lenses slow rather than merely delay myopia progression. This hypothesis predicts that during the first two years of the BLINK2 Study, when all subjects will wear soft bifocal contact lenses, subjects will progress at the same rate regardless of original lens assignment in the BLINK Study. Alternatively, faster myopia progression in subjects originally fitted with soft bifocal contact lenses compared to single vision contact lenses would indicate a delay in myopia progression rather than a permanent treatment benefit.
Rebound of progression | One year
  In the event of an effect of multifocal contact lens on myopia progression, the investigators will test the hypothesis that there is no increase in myopia when switching from bifocal to single vision contact lenses. This hypothesis predicts that the progression of myopia during the last year of follow-up when all subjects will switch to single vision contact lenses, will be similar to myopia progression during the first two years when all subjects wore bifocal contact lenses. Alternatively, faster progression after switching to single vision contact lens wear indicates a "rebound" of myopia progression.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Walline, OD PhD, Principal Investigator — The Ohio State University College of Optometry
Locations (2):
- United States (2):
  - Ohio State University, Columbus, Ohio
  - University of Houston, Houston, Texas

REFERENCES:
- [Derived] Chandler MA, Robich ML, Jordan LA, Mutti DO, Berntsen DA, Fenton R, Day E, Walline JJ; BLINK2 Study Group. Accommodation in Children after 4.7 Years of Multifocal Contact Lens Wear in the BLINK Study Randomized Clinical Trial. Optom Vis Sci. 2023 Jul 1;100(7):425-431. doi: 10.1097/OPX.0000000000002040. Epub 2023 Jun 24. PMID 37369096